CLINICAL TRIAL: NCT01423747
Title: Allogeneic Stem Cell Transplantation in Children and Adolescents With Acute Lymphoblastic Leukaemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Anna Kinderkrebsforschung (Other)
Collaborators: International BFM Study Group (Network)
Responsible Party: Principal Investigator, Prof. Christina Peters, MD, PHD, St. Anna Kinderspital, Austria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALL-SZT- BFM 2003
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood;
Keywords: ALL; HSCT; children; adolescents
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Etoposide; Whole-Body Irradiation; fludarabine; Muromonab-CD3; treosulfan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MSD - matched sibling donor (Other): patients with a MSD receive a conditioning of total body irradiation (TBI) (12 Gy, 6 fractions) and VP16 60mg/kg for one day (-3)
  Interventions: Drug: VP16; Radiation: TBI
- MD - matched donor (Other): patients with a HLA (Human Leukocyte Antigen) matched unrelated Donor (9/10 oder 10/10) receive total body irradiation (TBI) (12Gy in 6 fractions), VP16 60mg/kg/d on day -3 and ATG fresenius 20mg/kg/d on day -3,-2,-1
  Interventions: Drug: VP16, ATG; Radiation: TBI
- MMD - mismatched Donor (Other): Patients with a mismatched donor receive stem cells either from cord blood, a haploidentical donor (parent) or from a non-related donor with a match less or equal 8/10
  Interventions: Drug: Fludarabine, OKT3, Treosulfan, Thiotepa; Drug: VP16, ATG; Radiation: TBI

INTERVENTIONS:
Drug: VP16 — patients with MSD receive as conditioning VP16 60mg/kg/d on day -3
  Other Names: Etoposid
  Arms: MSD - matched sibling donor
Radiation: TBI — patients with a MSD receive TBI (12Gy in 6 fractions) as conditioning
  Other Names: total body irradiation
  Arms: MSD - matched sibling donor
Drug: VP16, ATG — patients with a HLA matched unrelated Donor (9/10 oder 10/10) receive VP16 60mg/kg/d on day -3 and ATG fresenius 20mg/kg/d on day -3,-2,-1
  Other Names: Etoposid, Antithymoglobuline
  Arms: MD - matched donor
Radiation: TBI — patients with a HLA matched unrelated Donor (9/10 oder 10/10) receive TBI (12Gy in 6 fractions)
  Other Names: total body irradiation
  Arms: MD - matched donor
Drug: Fludarabine, OKT3, Treosulfan, Thiotepa — patients with a MMD (haploidentical or cord blood) receive Fludarabine 30mg/m²/d on day -9 to -5, ATG 20mg/kd/d on day -3 to day -1, Treosulfan 14g/m²/d on day -7 to -5 and Thiotepa 2x5mg/kg/d on day -4
  Other Names: ATG:Antithymoglobuline
  Arms: MMD - mismatched Donor
Drug: VP16, ATG — patients with MMD-transplantation (8/10)receive VP16 60mg/kg/d on day -4, ATG from day -3 to day-1 20mg/kg/d
  Other Names: Etoposid, Antithymoglobuline
  Arms: MMD - mismatched Donor
Radiation: TBI — patients with a MMD-transplantation (8/10) receive 12 Gy in 6 fractions
  Other Names: total body irradiation
  Arms: MMD - mismatched Donor

SUMMARY:
With this protocol the ALL-SZT BFM international study group wants

to evaluate whether hematopoietic stem cell transplantation (HSCT) from matched family or unrelated matched donors (MD) is equivalent to the HSCT from matched sibling donors (MSD).

to evaluate the efficacy of haematopoietic stem cell transplantation (HSCT) from mismatched family or unrelated mismatched donors (MMD) as compared to HSCT from matched sibling donor (MSD) and matched donor (MD).

to determine whether therapy has been carried out according to the main haematopoietic stem cell transplantation (HSCT) protocol recommendations. The standardisation of the treatment options during haematopoietic stem cell transplantation (HSCT) from different donor types aims at the achievement of an optimal comparison of survival after HSCT with survival after chemotherapy only.

to prospectively evaluate and compare the incidence of acute and chronic graft- versus-host-disease (GvHD) after haematopoietic stem cell transplantation (HSCT) from matched sibling donor (MSD), from matched donor (MD) and from mismatched donor (MMD).

DETAILED DESCRIPTION:
Patients with high risk or relapsed acute lymphoblastic leukaemia (ALL) have a worse prognosis compared to all other patients with ALL. For these patients additional therapy approaches are required after they have achieved remission with multimodal chemotherapy. Allogeneic haematopoetic stem cell transplantation shows promising results mainly due to an immunological antileukaemic control by the graft-versus-leukaemia effect, but treatment related mortality and morbidity remains a serious problem.

ELIGIBILITY:
Inclusion Criteria:

* age at time of initial diagnosis or relapse diagnosis, respectively under or equal 18 years
* indication for allogeneic hematopoietic stem cell transplantation (HSCT)
* complete remission before hematopoietic stem cell transplantation (HSCT)
* written consent of the parents (legal guardian) and, if necessary, the minor patient via Informed Consent Form
* no pregnancy
* no secondary malignancy
* no previous hematopoietic stem cell transplantation (HSCT)
* hematopoietic stem cell transplantation (HSCT) is performed in a study participating centre.

Exclusion Criteria:

* age at time of initial diagnosis or relapse diagnosis, respectively above 18 years
* no indication for allogeneic HSCT
* no complete remission before SCT
* no written consent of the parents (legal guardian) and, if necessary, the minor patient via Informed Consent Form
* pregnancy
* secondary malignancy
* previous HSCT
* HSCT is not performed in a study participating centre.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2003-07; Primary Completion 2011-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Event-free and overall survival after allogeneic haematopoietic stem cell transplantation (HSCT) | 14 years

SECONDARY OUTCOMES:
occurrence of acute and chronic Graft-versus-Host-Disease (GvHD) | 14 years
  Evaluation of the incidence and severity of acute Grade I-IV Graft-versus-Host-Disease (GvHD) and of limited or extensive chronic GvHD
occurrence and course of late effects after chemotherapy with subsequent allogeneic hematopoietic stem cell transplantation (HSCT) | 14 years
  valuation of organ dysfunctions according to WHO Toxicity score
occurrence and course of late effects after chemotherapy with subsequent allogeneic hematopoietic stem cell transplantation (HSCT) | 14
  evaluation of growth retardation and endocrine dysfunction
occurrence and course of late effects after chemotherapy with subsequent allogeneic hematopoietic stem cell transplantation (HSCT) | 14 years
  Evaluation of incidence of aseptic bone necrosis
occurrence and course of secondary malignancies after chemotherapy with subsequent allogeneic hematopoietic stem cell transplantation (HSCT) | 14 years
  Evaluation of incidence of secondary cancer after total body irradiation (TBI) and/or chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Arend v. Stackelberg, MD, PhD, Study Chair — ALL-REZ BFM Study Center Berlin Germany; Martin Schrappe, MD, Prof., Study Chair — ALL BFM study center Kiel, Germany
Locations (24):
- Austria (3):
  - Universitätsklinik für Kinder- und Jugendheilkunde, Klin. Abt. f. Hämato-Onkologie, Graz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Innsbruck
  - St. Anna Kinderspital, Vienna
- Germany (21):
  - Charité Campus Virchow- Klinikum, Klinikum der Pädiatrie, Onkologie/Hämatologie/KMT, Berlin
  - Klinik und Poliklinik für Kinderheilkunde, Hämatologie, Onkologie, Dresden
  - Universitätsklinikum Düsseldorf, Klinik f. Kinderonkologie, Hämatologie u. Immunologie, Düsseldorf
  - Klinik für Kinder und Jugendliche der Universität Erlangen-Nürnberg, Erlangen
  - Universitätsklinikum Essen, Zentrum für Kinderheilkunde, Abt. für Hämatologie/Onkologie, Essen
  - Klinik für Kinderheilkunde III, Hämatologie und Onkologie, Johann Wolfgang Goethe Universität, Frankfurt am Main
  - Universitätsklinikum Freiburg, Zentrum für Kinderheilkunde und Jugendmedizin, Klinik IV: Päd. Hämatologie und Onkologie, Freiburg im Breisgau
  - Zentrum für Kinderheilkunde, Abt. Hämatologie und Onkologie, Giessen
  - Klinkum der Med. Fakultät der Martin-Luther-Universität Halle-Wittenberg, Uni. Klinik un Poliklinik für Kinder- und Jugendmedizin, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Kinderklinik, Abt. für Hämatologie und Onkologie, Hamburg
  - Med. Hochschule Hannover, Päd. Hämatologie und Onkologie, Hanover
  - Universitätskinderklinik, Päd. Hämatologie, Onkologie und Immunologie, Heidelberg
  - Klinik für Knochenmarktransplantation, Idar-Oberstein
  - Klinik für Kinder- und Jugendmedizin, Jena
  - Universitätsklinikum Kiel, Klinik für Allgemeine Pädiatrie, Kiel
  - Klinikum der Universität München, Dr. von Haunersches Kinderspital, Abt. für Hämatologie / Onkologie, München
  - Städt. Krankenhaus München-Schwabing, Universitätskinderklinik der TU, München
  - Universitätsklinikum Münster, Klinik und Poliklinik für Kinderheilkunde, päd. Hämatologie / Onkologie, Münster
  - Univ.-Klinik für Kinderheilkunde und Jugendmedizin, Tübingen
  - Universitätskinderklinik, Ulm
  - Universitätsklinik, päd. Onkologie/Stammzelltransplantation, Würzburg

REFERENCES:
- [Result] Peters C, Schrauder A, Schrappe M, von Stackelberg A, Stary J, Yaniv I, Gadner H, Klingebiel T; BFM Study Group, the IBFM-Study Group and the Paediatric Disease Working Party of the EBMT. Allogeneic haematopoietic stem cell transplantation in children with acute lymphoblastic leukaemia: the BFM/IBFM/EBMT concepts. Bone Marrow Transplant. 2005 Mar;35 Suppl 1:S9-11. doi: 10.1038/sj.bmt.1704835. PMID 15812540
- [Result] Pulsipher MA, Peters C, Pui CH. High-risk pediatric acute lymphoblastic leukemia: to transplant or not to transplant? Biol Blood Marrow Transplant. 2011 Jan;17(1 Suppl):S137-48. doi: 10.1016/j.bbmt.2010.10.005. PMID 21195303
- [Result] Peters C, Schrappe M, von Stackelberg A, Schrauder A, Bader P, Ebell W, Lang P, Sykora KW, Schrum J, Kremens B, Ehlert K, Albert MH, Meisel R, Matthes-Martin S, Gungor T, Holter W, Strahm B, Gruhn B, Schulz A, Woessmann W, Poetschger U, Zimmermann M, Klingebiel T. Stem-cell transplantation in children with acute lymphoblastic leukemia: A prospective international multicenter trial comparing sibling donors with matched unrelated donors-The ALL-SCT-BFM-2003 trial. J Clin Oncol. 2015 Apr 10;33(11):1265-74. doi: 10.1200/JCO.2014.58.9747. Epub 2015 Mar 9. PMID 25753432
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441
- [Derived] Preuner S, Peters C, Potschger U, Daxberger H, Fritsch G, Geyeregger R, Schrauder A, von Stackelberg A, Schrappe M, Bader P, Ebell W, Eckert C, Lang P, Sykora KW, Schrum J, Kremens B, Ehlert K, Albert MH, Meisel R, Lawitschka A, Mann G, Panzer-Grumayer R, Gungor T, Holter W, Strahm B, Gruhn B, Schulz A, Woessmann W, Lion T. Risk assessment of relapse by lineage-specific monitoring of chimerism in children undergoing allogeneic stem cell transplantation for acute lymphoblastic leukemia. Haematologica. 2016 Jun;101(6):741-6. doi: 10.3324/haematol.2015.135137. Epub 2016 Feb 11. PMID 26869631
- [Derived] Bader P, Kreyenberg H, von Stackelberg A, Eckert C, Salzmann-Manrique E, Meisel R, Poetschger U, Stachel D, Schrappe M, Alten J, Schrauder A, Schulz A, Lang P, Muller I, Albert MH, Willasch AM, Klingebiel TE, Peters C. Monitoring of minimal residual disease after allogeneic stem-cell transplantation in relapsed childhood acute lymphoblastic leukemia allows for the identification of impending relapse: results of the ALL-BFM-SCT 2003 trial. J Clin Oncol. 2015 Apr 10;33(11):1275-84. doi: 10.1200/JCO.2014.58.4631. Epub 2015 Jan 20. PMID 25605857